CLINICAL TRIAL: NCT00106574
Title: A Randomized, Double-blind Study of the Effect of Tocilizumab on Reduction in Signs and Symptoms in Patients With Moderate to Severe Active Rheumatoid Arthritis and Inadequate Response to DMARD Therapy
Brief Title: A Study to Assess the Effect of Tocilizumab + DMARD Therapy on Signs and Symptoms in Patients With Moderate to Severe Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA18063
Record Dates: First submitted 2005-03-25; First posted 2005-03-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — iv every 4 weeks
  Arms: 2
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks
  Arms: 1

SUMMARY:
This 2 arm study will compare the safety and efficacy, with regard to reduction of signs and symptoms, of tocilizumab versus placebo in combination with traditional Disease-Modifying Anti-Rheumatic Drug (DMARD) therapy in patients with moderate to severe active rheumatoid arthritis (RA) who have had an inadequate response to current DMARD therapy. Patients will be randomized to receive tocilizumab 8mg/kg iv or placebo iv every 4 weeks, in conjunction with stable DMARD therapy. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients at least 18 years of age with moderate to severe active RA for at least 6 months;
* inadequate response to current anti-rheumatic therapies, including 1 or more traditional DMARDs;
* stable DMARD therapy for at least 8 weeks before entering study;
* patients of reproductive potential must be using reliable methods of contraception.

Exclusion Criteria:

* major surgery (including joint surgery) within 8 weeks before entering study, or planned surgery within 6 months after entering study;
* patients who have previously failed treatment with an anti-tumor necrosis factor agent;
* women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ACR 20 response | Week 24

SECONDARY OUTCOMES:
Percentage of patients with ACR 50 and ACR 70 responses. | Week 24
Mean changes in parameters of ACR core set | Week 24
AEs, laboratory parameters, vital signs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (134):
- United States (74):
  - Mesa, Arizona
  - Paradise Valley, Arizona
  - Peoria, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Palm Desert, California
  - Palo Alto, California
  - San Jose, California
  - Upland, California
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Delray Beach, Florida
  - Jupiter, Florida
  - Palm Habor, Florida
  - Palm Harbor, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Springfield, Illinois
  - Vernon Hills, Illinois
  - Indianapolis, Indiana
  - Bowling Green, Kentucky
  - Baton Rouge, Louisiana
  - Shreverport, Louisiana
  - Frederick, Maryland
  - Boston, Massachusetts
  - Lansing, Michigan
  - Duluth, Minnesota
  - Eagan, Minnesota
  - Saint Louis Park, Minnesota
  - Springfield, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Reno, Nevada
  - Clifton, New Jersey
  - Haddon Heights, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Plainview, New York
  - Roslyn, New York
  - Smithtown, New York
  - Syracuse, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Gallipolis, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Rockledge, Pennsylvania
  - Willow Grove, Pennsylvania
  - Johnston, Rhode Island
  - Charleston, South Carolina
  - Hixson, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Mesquite, Texas
  - Burlington, Vermont
  - Arlington, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Vancouver, Washington
  - La Crosse, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Rosario
- Australia (2):
  - Parkville
  - Sydney
- Brazil (3):
  - Campinas
  - Goiânia
  - Rio de Janeiro
- Canada (5):
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- China (2):
  - Beijing
  - Shanghai
- San José, Costa Rica
- Czechia (2):
  - Hradec Králové
  - Prague
- Finland (2):
  - Helsinki
  - Jyväskylä
- France (12):
  - Boulogne-Billancourt
  - Clermont-Ferrand
  - Grenoble
  - Limoges
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Pierre-Bénite
  - Rennes
  - Saint-Etienne
  - Tours
- Germany (7):
  - Aachen
  - Essen
  - Hildesheim
  - München
  - Osnabrück
  - Sendenhorst
  - Stuttgart
- Hong Kong (2):
  - Hong Kong
  - Tuenmen
- Mexico (3):
  - León
  - Mexico City
  - Tijuana
- Panama City, Panama
- Russia (4):
  - Moscow
  - Ryazan
  - Saint Petersburg
  - Tula
- South Africa (3):
  - Durban
  - Pretoria
  - Radiokop
- Spain (5):
  - Barakaldo
  - Madrid
  - Málaga
  - Pontevedra
  - Santiago de Compostela
- Sweden (2):
  - Stockholm
  - Umeå
- Thailand (2):
  - Bangkok
  - Chiang Mai

REFERENCES:
- [Derived] Welsh P, Tuckwell K, McInnes IB, Sattar N. Effect of IL-6 receptor blockade on high-sensitivity troponin T and NT-proBNP in rheumatoid arthritis. Atherosclerosis. 2016 Nov;254:167-171. doi: 10.1016/j.atherosclerosis.2016.10.016. Epub 2016 Oct 8. PMID 27744141
- [Derived] Keystone EC, Anisfeld A, Ogale S, Devenport JN, Curtis JR. Continued benefit of tocilizumab plus disease-modifying antirheumatic drug therapy in patients with rheumatoid arthritis and inadequate clinical responses by week 8 of treatment. J Rheumatol. 2014 Feb;41(2):216-26. doi: 10.3899/jrheum.130489. Epub 2014 Jan 15. PMID 24429164
- [Derived] Wang J, Bansal AT, Martin M, Germer S, Benayed R, Essioux L, Lee JS, Begovich A, Hemmings A, Kenwright A, Taylor KE, Upmanyu R, Cutler P, Harari O, Marchini J, Criswell LA, Platt A. Genome-wide association analysis implicates the involvement of eight loci with response to tocilizumab for the treatment of rheumatoid arthritis. Pharmacogenomics J. 2013 Jun;13(3):235-41. doi: 10.1038/tpj.2012.8. Epub 2012 Apr 10. PMID 22491018
- [Derived] Genovese MC, McKay JD, Nasonov EL, Mysler EF, da Silva NA, Alecock E, Woodworth T, Gomez-Reino JJ. Interleukin-6 receptor inhibition with tocilizumab reduces disease activity in rheumatoid arthritis with inadequate response to disease-modifying antirheumatic drugs: the tocilizumab in combination with traditional disease-modifying antirheumatic drug therapy study. Arthritis Rheum. 2008 Oct;58(10):2968-80. doi: 10.1002/art.23940. PMID 18821691